CLINICAL TRIAL: NCT07387978
Title: A Pilot Study to Describe the Effect of Photobiomodulation in Reducing the Severity and Incidence of Oral Mucositis in Oral Cancer Patients Undergoing Radiation Treatment
Brief Title: A Study to Describe the Effect of Photobiomodulation (Low Level Laser Therapy) in Reducing the Severity and Incidence of Oral Mucositis (Oral Ulceration) in Oral Cancer Patients Undergoing Radiation Treatment
Acronym: PBM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25/131
Record Dates: First submitted 2025-12-17; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Oral Mucositis
Keywords: photobiomodulation; low level laser therapy; head and neck cancer; oral cancer; radiotherapy; oral mucositis
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms; Mouth Neoplasms | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Photobiomodulation (Experimental): Participants will receive photobiomodulation therapy five times a week during the course of their radiation treatment. Upon completion of radiotherapy, if oral mucositis is still present, participants can choose to continue photobiomodulation treatment until oral mucositis has resolved. The frequency of photobiomodulation will be conducted at the discretion of the investigator.
  Interventions: Device: photobiomodulation

INTERVENTIONS:
Device: photobiomodulation — photobiomodulation (low level laser therapy) application within and outside the oral cavity

SUMMARY:
The goal of this study is to describe the effect of photobiomodulation (PBM) on the incidence and severity of oral mucositis in post-operative oral cancer patients receiving radiotherapy +/- chemotherapy.

Participants will receive PBM treatment five times a week throughout the course of their radiotherapy.

The main question it aims to answer is whether photobiomodulation reduces the incidence and severity of oral mucositis.

DETAILED DESCRIPTION:
BACKGROUND: Strong evidence exists within the literature regarding the effectiveness and safety of PBM in preventing oral mucositis in head and neck cancer patients. PBM is recommended in the Multinational Association of Supportive Care in Cancer and National Institute of Health and Care Excellence oral mucositis prevention guidelines, as a treatment modality for oral mucositis prevention in H&N cancer patients. PBM using the THOR laser has received TGA approval for use in prevention and treatment of oral mucositis in Australia.

PARTICIPANTS: post operative oral cancer patients, with clear margins, planned for radiotherapy (50Gy or greater) +/- chemotherapy.

METHODS: participants will receive PBM treatment five times a week throughout the course of their radiotherapy.

EXPECTED OUTCOMES: decrease in incidence and severity of oral mucositis, decrease in pain levels and improved quality of life, less need for analgesia, increased ability to maintain oral intake, less severe trismus, lower rates of hospitalization

ELIGIBILITY:
Inclusion Criteria:

* Patient has provided written informed consent using the PBM PICF
* Age ≥ 18 years of age at Screening
* Histological diagnosis of HNC of the oral cavity with no evidence of macroscopic or microscopic residual disease post-surgery (R0 or R1 resection) with histopathological confirmation and no gross residual lymphadenopathy in the planned PBM treatment area
* Planned treatment with RT or chemoradiotherapy to a dose of ≥ 50 Gy Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 (Appendix 1)
* Intact oral mucosa (no visible ulceration, dehiscence, or active infection)

Exclusion Criteria:

* Gross macroscopic and/or microscopic residual disease post-surgery (R2 resection) or gross residual lymphadenopathy in the planned PBM treatment area
* Prior RT to the head and neck including the oral or oropharyngeal mucosa
* Prior cytotoxic chemotherapy in the last 3 months
* Diagnosis of photosensitive disorder (cutaneous porphyria, xeroderma pigmentosum, etc)
* Concurrent administration of cetuximab
* Known to be pregnant or planning to become pregnant within the trial period
* Diagnosis of epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence and severity of acute oral mucositis | Through study completion, an average of 1 year
  To describe the effect of PBM on the cumulative incidence and severity of acute OM as defined by the Common Terminology Criteria for Adverse Events, version 5.0 (CTCAE v5.0) for radiation induced mucositis during RT and for 8 weeks following RT.

SECONDARY OUTCOMES:
Function and quality of life (QoL) | Through study completion, an average of 1 year
  Quantitative analysis of MD Anderson Symptom Inventory for Head and Neck Cancer scores to describe the effect of PBM on function and QoL
Pain in the oral cavity and throat | Through study completion, an average of 1 year
  Quantitative analysis of Oral Mucositis Weekly Questionnaire-Head and Neck scores to describe effect of PBM on oral cavity and throat pain
Analgesia intake | Through study completion, an average of 1 year
  Concurrent use of analgesic medications and mouthwashes to determine effect of PBM on need for analgesia (yes/no)
Need for enteral feeding | Through study completion, an average of 1 year
  Use of enteral feeding to describe effect of PBM on ability to maintain oral intake
Hospitalisation rates | Through study completion, an average of 1 year
  Hospitalisation rates due to mucositis in the oral cavity or related events will be documented
Trismus | Through study completion, an average of 1 year
  Maximal-interincisal opening. For participants who are edentulous, the distance from the edentulous ridge to the opposing side vertically will be used instead

CONTACTS AND LOCATIONS:
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
This is a single institution study

REFERENCES:
- [Background] Bensadoun, R. J., Epstein, J. B., Nair, R. G., Barasch, A., Raber-Durlacher, J. E., Migliorati, C., Genot-Klastersky, M. T., Treister, N., Arany, P., & Lodewijckx, J. (2020). Safety and efficacy of photobiomodulation therapy in oncology: A systematic review. Cancer medicine, 9(22), 8279-8300. Brandão, T. B., Morais-Faria, K., Ribeiro, A. C. P., Rivera, C., Salvajoli, J. V., Lopes, M. A., Epstein, J. B., Arany, P. R., de Castro, G., & Migliorati, C. A. (2018). Locally advanced oral squamous cell carcinoma patients treated with photobiomodulation for prevention of oral mucositis: retrospective outcomes and safety analyses. Supportive Care in Cancer, 26, 2417-2423. Courtois, E., Bouleftour, W., Guy, J. B., Louati, S., Bensadoun, R. J., Rodriguez-Lafrasse, C., & Magné, N. (2021). Mechanisms of PhotoBioModulation (PBM) focused on oral mucositis prevention and treatment: a scoping review. BMC Oral Health, 21(1), 220. Elad, S., Cheng, K. K. F., Lalla, R. V., Yarom, N., Hong, C., Logan, R. M., Bowen, J., Gibson, R., Saunders, D. P., & Zadik, Y. (2020). MASCC/ISOO clinical practice guidelines for the management of mucositis secondary to cancer therapy. Cancer, 126(19), 4423-4431. Macann, A., Fua, T., Milross, C. G., Porceddu, S. V., Penniment, M., Wratten, C., Krawitz, H., Poulsen, M., Tang, C. I., & Morton, R. P. (2014). Phase 3 trial of domiciliary humidification to mitigate acute mucosal toxicity during radiation therapy for head-and-neck cancer: first report of Trans Tasman Radiation Oncology Group (TROG) 07.03 RadioHUM study. International Journal of Radiation Oncology* Biology* Physics, 88(3), 572-579. NICE. (2018). Low-level laser therapy for preventing or treating oral mucositis caused by radiotherapy or chemotherapy. Sroussi, H. Y., Epstein, J. B., Bensadoun, R. J., Saunders, D. P., Lalla, R. V., Migliorati, C. A., Heaivilin, N., & Zumsteg, Z. S. (2017). Common oral complications of head and neck cancer radiation therapy: mucositis, infections, saliva cha
- [Background] Taylor, J. K.-A., Mady, L. J., Baddour, K., Iheagwara, U. K., Zhai, S., Ohr, J. P., Zandberg, D. P., Gorantla, V. C., Ferris, R. L., & Kim, S. (2022). A phase Ⅱ prospective trial of photobiomodulation therapy in limiting oral mucositis in the treatment of locally advanced head and neck cancer patients. World Journal of Otorhinolaryngology-Head and Neck Surgery, 8(04), 345-354.
- [Background] Sroussi, H. Y., Epstein, J. B., Bensadoun, R. J., Saunders, D. P., Lalla, R. V., Migliorati, C. A., Heaivilin, N., & Zumsteg, Z. S. (2017). Common oral complications of head and neck cancer radiation therapy: mucositis, infections, saliva change, fibrosis, sensory dysfunctions, dental caries, periodontal disease, and osteoradionecrosis. Cancer medicine, 6(12), 2918-2931
- [Background] NICE. (2018). Low-level laser therapy for preventing or treating oral mucositis caused by radiotherapy or chemotherapy.
- [Background] Macann, A., Fua, T., Milross, C. G., Porceddu, S. V., Penniment, M., Wratten, C., Krawitz, H., Poulsen, M., Tang, C. I., & Morton, R. P. (2014). Phase 3 trial of domiciliary humidification to mitigate acute mucosal toxicity during radiation therapy for head-and-neck cancer: first report of Trans Tasman Radiation Oncology Group (TROG) 07.03 RadioHUM study. International Journal of Radiation Oncology* Biology* Physics, 88(3), 572-579
- [Background] Elad, S., Cheng, K. K. F., Lalla, R. V., Yarom, N., Hong, C., Logan, R. M., Bowen, J., Gibson, R., Saunders, D. P., & Zadik, Y. (2020). MASCC/ISOO clinical practice guidelines for the management of mucositis secondary to cancer therapy. Cancer, 126(19), 4423-4431.
- [Background] Courtois, E., Bouleftour, W., Guy, J. B., Louati, S., Bensadoun, R. J., Rodriguez-Lafrasse, C., & Magné, N. (2021). Mechanisms of PhotoBioModulation (PBM) focused on oral mucositis prevention and treatment: a scoping review. BMC Oral Health, 21(1), 220.
- [Background] Brandão, T. B., Morais-Faria, K., Ribeiro, A. C. P., Rivera, C., Salvajoli, J. V., Lopes, M. A., Epstein, J. B., Arany, P. R., de Castro, G., & Migliorati, C. A. (2018). Locally advanced oral squamous cell carcinoma patients treated with photobiomodulation for prevention of oral mucositis: retrospective outcomes and safety analyses. Supportive Care in Cancer, 26, 2417-2423.
- [Background] Bensadoun, R. J., Epstein, J. B., Nair, R. G., Barasch, A., Raber-Durlacher, J. E., Migliorati, C., Genot-Klastersky, M. T., Treister, N., Arany, P., & Lodewijckx, J. (2020). Safety and efficacy of photobiomodulation therapy in oncology: A systematic review. Cancer medicine, 9(22), 8279-8300.